CLINICAL TRIAL: NCT00176592
Title: Phase IV, Rater-blinded, Randomized Study, Comparing 250 mg of Betaseron With 20 mg of Copaxone in Patients With the Relapsing-remitting(RR) or CIS Forms of ms Using 3 Tesla(3T) Magnetic Resonance Imaging (MRI) With Triple-dose Gadolinium
Brief Title: Phase IV Study, Betaseron Versus Copaxone for Relapsing Remitting or CIS Forms of MS Using Triple Dose Gad 3 T MRI
Acronym: BECOME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Principal Investigator, Suhayl Dhib-Jalbut, MD, Professor and Chair, Department of Neurology, NJMS & RWJMS, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0120020167; 0120020167 (Other: Rutgers)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Brain; Betaseron; Copaxone; MRI
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betaseron (Active Comparator): Betaseron 250 micrograms SQ every other day and Triple-Dose Gadolinium at each MRI
  Interventions: Drug: Betaseron
- Copaxone (Active Comparator): Copaxone 20 mg daily SQ and Triple-Dose Gadolinium at each MRI
  Interventions: Drug: Copaxone

INTERVENTIONS:
Drug: Betaseron — Betaseron 250 micrograms injected SQ every other day
  Other Names: Betaseron 250 mcg SQ every other day; Intaferon beta 1 b
  Arms: Betaseron
Drug: Copaxone — Copaxone 20 mg injected SQ every day (glatiramer acetate)
  Other Names: Copaxone 20 mg injected SQ every day (glatiramer acetate)
  Arms: Copaxone

SUMMARY:
This is the first comparison of efficacy of Betaseron and Copaxone for treatment of relapsing forms of MS.

DETAILED DESCRIPTION:
We propose to perform a head to head comparison of Interferon beta and Copaxone for treatment of patients with CIS and RR forms of MS using acute changes on MRI as primary outcome. The study will be performed at the two clinical practice sites of the Multiple Sclerosis Center at University of Medicine and Dentistry New Jersey-New Jersey Medical School, One of the two FDA approved preparations of higher dose interferon beta (Betaseron) will be compared at standard dose every other day (QOD) 250 ug subcutaneously(SQ) with Copaxone at 20mg SQ daily (QD) in 70 to 80 patients. Although the current approved plan is to perform monthly MRIs for 1 year followed by another MRI at 2 years, the protocol has been changed to continue performing monthly MRIs during the second year of the study for all patients who complete their first year and up to January 31, 2006 when the study will end. The study uses brain imaging with 3 Tesla MRI with triple dose Gadolinium for primary and secondary outcomes and several clinical and cognitive measures for secondary outcomes. The sample size was estimated to detect a 40-50% difference in the number of active MS lesions by MRI between the two arms at 1 year follow up, consistent with the primary outcome measure. The primary outcome measure is the number of "combined-active" lesions by monthly MRI at the conclusion of the study, which includes contrast enhancing lesions and non-enhancing lesions on long Time repetition (TR) scans that have appeared since the most recent examination. Several secondary MRI outcome measures are studied in addition to the number of enhancing lesions and the number of new lesions on long TR images. We will examine the number of patients who remain "combined-active disease-free" for the duration of the study and the number of "combined-active disease-free" scans. Apart from these traditional methods of analysis by a reader who will be blinded to patient clinical status and therapy, objective volumetric analysis will be carried out. Making use of both automated and manual techniques, we will determine the overall burden of disease (the volume of lesions on long TR scans), the burden of active disease (the volume of brain enhancement) and the burden of chronic disease (the volume of lesions that are markedly hypointense on T1). Another MRI outcome measures will be detection of diffusion anisotropy differences, MR spectroscopy, and magnetization transfer ratio as summarized in Appendix 5. These new techniques have shown promise for detecting disease that cannot be detected with conventional MRI (13, 37).

In addition to MRI, several clinical and cognitive outcome measures will be used for secondary analysis. These include the number and severity of relapses measured by different methods, and change in disability measured by the Expanded Disability Status Scale (EDSS), the Neurological Rating Scale, and the Multiple Sclerosis Functional Composite (MSFC). The cognitive measures will be the subject's neurocognitive function measured by standard neurocognitive examination obtained by a licensed neuropsychologist and the Cognitive Stability Index (CSI), a novel Internet-based test of cognitive function in addition to the Paced Auditory Serial Addition Test (PASAT),which is a component of the MSFC.

ELIGIBILITY:
Inclusion criteria:

Patients must meet all of the following criteria at the time of the baseline visit in order to enter the trial:

* Be Between 18 and 55 years of age, at baseline.
* Be capable of informed consent in English prior to any study related procedures.Spanish speaking patients who do not read English well can give written informed consent if a relative or friend fluent in both English and Spanish has translated the consent and any questions the patient may have.
* Be available and willing to complete all study assessments.
* Presently meet one of the two following forms of multiple sclerosis:

  1. Relapsing-remitting ms plus evidence of recent disease activity as shown by the development of one or more clinical and/or MRI lesions during the 6 months prior to entry into the study.
  2. A CIS consistent with central nervous system (CNS) demyelination confirmed on ophthalmologic or neurological examination with onset within 6 months prior to study entry. Also:a- evidence of dissemination in space, there should be two or more brain MRI lesions ≥ 3 mm in size at least one of which should be ovoid and/or periventricular in location; and b- As evidence of dissemination in time, if the CIS is acute (≤1 month) there should be one or more non-enhancing lesion or if the CIS is not acute (older than 1 month) the MRI should show one or more enhancing lesions.

     * At baseline, have an EDSS between 0-5.5.
* Females of childbearing potential must agree to practice adequate contraception methods. All females must have negative pregnancy test results at screening and a negative urine pregnancy test at baseline.
* Screening laboratory results that confirm adequate bone marrow, renal, and hepatic function.

Exclusion criteria

Patients were not permitted into the study if they met any of the following criteria:

* Onset of a relapse between screening and Study Day 1.
* Present evidence or history of any conditions that could affect the CNS or interfere with the MRI results or any other evaluation in the study.
* Possess any of the standard metallic devices or foreign bodies that are contraindications for MRI.
* Patient weight and or size unable to fit in the 3T MRI scanner.
* Pregnancy, as denoted by a positive serum pregnancy test at screening visit or a positive urine pregnancy test at the baseline visit. Subjects who are breast-feeding are also excluded.
* Have a known allergy or hypersensitivity to Gadolinium-chelates, human proteins including albumin and interferons, or Glatiramer Acetate or Mannitol.
* Uncontrolled, clinically significant heart diseases, such as dysrhythmias, angina, or uncompensated congestive heart failure. History of or current unstable medical conditions that could be deemed clinically significant.
* Intolerance or any contraindication to acetaminophen, ibuprofen, or steroids.
* Inability, in the opinion of the principal investigator or staff, to be compliant with protocol requirements for the duration of the study.
* Participation in any clinical trial within the past six months
* History or present evidence of addictions.
* Have active peptic ulcer disease.
* Inability to have subcutaneous injections administered.
* Medical, psychiatric or other conditions that compromise the patient's ability to understand the study procedures.
* Claustrophobia.
* Uncontrolled head movements.
* Treatment with any of the following in the indicated time frames: Any of the Interferons for > 6 months· Glatiramer acetate (Copaxone) for > 6 months.No prior use allowed of Total lymphoid irradiation, Anti-lymphocyte monoclonal antibody (e.g.(Campath-1H) .Mitoxantrone,cyclophosphamide, Azathioprine, intravenous immunoglobulin (IVIG), cyclosporine within 6 months before the screening visit·Any investigational drug 21 days before screening visit·Systemic corticosteroids·ACTH from screening visit through Study Day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2003-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Cook, MD, Principal Investigator — MD
Locations (1):
- New Jersey Medical School, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cadavid D, Wolansky LJ, Skurnick J, Lincoln J, Cheriyan J, Szczepanowski K, Kamin SS, Pachner AR, Halper J, Cook SD. Efficacy of treatment of MS with IFNbeta-1b or glatiramer acetate by monthly brain MRI in the BECOME study. Neurology. 2009 Jun 9;72(23):1976-83. doi: 10.1212/01.wnl.0000345970.73354.17. Epub 2009 Mar 11. PMID 19279320
- [Result] Cadavid D, Cheriyan J, Skurnick J, Lincoln JA, Wolansky LJ, Cook SD. New acute and chronic black holes in patients with multiple sclerosis randomised to interferon beta-1b or glatiramer acetate. J Neurol Neurosurg Psychiatry. 2009 Dec;80(12):1337-43. doi: 10.1136/jnnp.2008.171090. Epub 2009 Aug 16. PMID 19687024
- [Derived] Maranzano J, Rudko DA, Nakamura K, Cook S, Cadavid D, Wolansky L, Arnold DL, Narayanan S. MRI evidence of acute inflammation in leukocortical lesions of patients with early multiple sclerosis. Neurology. 2017 Aug 15;89(7):714-721. doi: 10.1212/WNL.0000000000004227. Epub 2017 Jul 19. PMID 28724581

RESULTS

PARTICIPANT FLOW:
Groups:
- Betaseron: Betaseron 250 micrograms SQ every other day
  Betaseron: Betaseron 250 micrograms injected SQ every other day
- Copaxone: 20 mg daily SQ
  Copaxone: Copaxone 20 mg injected SQ every day (glatiramer acetate)
Period: Overall Study
Arm/Group | Betaseron | Copaxone
Started | 36 | 39
Followed for 1 Year | 35 | 35
Followed for 2 Years | 29 | 35
Completed | 36 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Betaseron | Copaxone | Total
Number analyzed (Participants) | 36 | 39 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 39 | 75
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 36 [18 to 49] | 36 [22 to 55] | 36 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 9 | 14 | 23
Region of Enrollment [Number; unit: participants]
  United States | 36 | 39 | 75

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is the Number of "Combined Active Lesions" (CAL) by Monthly MRI at the Conclusion of the Study.
Description: Results are per patient mean number of lesions per scan. Results are per patient mean number of lesions per elapsed month. Contrasts types are: IFN 1b interferon beta 1b and GA glatiramer acetate.
Time Frame: up to 2 years
Population: Randomization was stratified by the presence or absence of enhancement. Analysis was intention to treat.
Measure: Mean (Standard Deviation); unit: Average number of lesions per scan
Units Other Than Participants: Combined Active Lesions
Arm/Group | Betaseron | Copaxone
Number analyzed (Participants) | 36 | 39
Number analyzed (Combined Active Lesions) | 1688 | 1053
Average number of lesions per scan | 0.63 (2.76) | 0.58 (2.46)
Statistical Analysis 1: Comparison: Betaseron vs Copaxone; This includes p value for rank sum test treatment comparison. This includes p value for rank sum test treatment comparison of intention to treat study population; Test type: Superiority — This includes p value for rank sum test treatment comparison. This includes p value for rank sum test treatment comparison of intention to treat study population; p < 0.05, Fisher Exact; Mean Difference (Final Values) = 0.05

2. Secondary Outcome: The Number of Enhancing Lesions.
Description: The first part of the secondary outcome measure is the total number of enhancing lesions per patient per treatment arm.
  The second part of the secondary outcome is the total number of new enhancing lesions per patient per treatment arm.
Time Frame: up to 2 years
Measure: Number; unit: New Enhancing Lesion
Units Other Than Participants: Enhancing Lesion
Arm/Group | Betaseron | Copaxone
Number analyzed (Participants) | 31 | 30
Number analyzed (Enhancing Lesion) | 1531 | 973
New Enhancing Lesion | 878 | 626

3. Secondary Outcome: The Number of MRI Disease Free Patients.
Description: The 1 year MRI results were used to determine the quantity of disease free patients per contrast type.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Betaseron | Copaxone
Number analyzed (Participants) | 36 | 39
participants
  The number of relapse-free patients at the completion of the study. | 19 | 28
  Free of combined active lesions, namely the combination of enhancing lesions plus new T2 lesions. | 7 | 10

ADVERSE EVENTS:
Time Frame: Adverse events in the form of symptoms were gathered over the duration of the study (24 months).
Description: Adverse events were recorded spontaneously and upon questioning by nurse at MRI for the hour of the MRI.
  Additional events were recorded at follow up visit within three months of MRI. Additional lab results were studied at follow up visit within three months of MRI.
  Finally, lab results and clinical adverse events were studied at three interim analyses by data monitoring committee.
Arm/Group | Betaseron | Copaxone
Serious Adverse Events (participants affected / at risk) | 7/36 | 7/39
Other Adverse Events (participants affected / at risk) | 2/36 | 7/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betaseron (N=36) | Copaxone (N=39)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) — One Patient had normal pregnancy and delivery. Discontinued drug and no longer participated in the study. Other two patients terminated pregnancy.
Malignant Nodule in Lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient had a chest x-ray that showed nodule which was malignant. Patient had surgery to remove 1 lobe, right lung.
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient experienced vomiting up all food and liquids; vertigo; severe gastroenteritis.
Loss of Hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Loss of hearing in left ear. Viral etiology. Treated by ENT.
Pain near IV Site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — During MRI, pain near IV site (right forearm). Extravasated contrast/IV fluid.Swelling, decreased skin temp, increased paresthesias and skin turned black near site.
Myelitis (Nervous system disorders) | 0 (0) | 1 (1) — Severe myelitis, bilateral leg weakness, dysesthesias, impaired balance.
Venous Thromboembolism (Blood and lymphatic system disorders) | 0 (0) | 1 (2) — Pain behind right knee while walking and standing. Deep vein thrombosis and pulmonary embolism. Treated at hospital.
Balance Impairment (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Patient experienced balance impairment for about 1 week; MRI showed multiple enhancing lesions.
Aneurysm (Vascular disorders) | 1 (1) | 0 (0) — Patient found to have three aneurysms. Two were clipped and one wrapped, Mild left sided stroke suffered.
Pancreatitis (Endocrine disorders) | 1 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Gastritis; nausea and vomiting; brainstem MS relapse.
Pain (General disorders) | 1 (1) | 0 (0) — Pain in right shoulder and leg. No foot sensation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betaseron (N=36) | Copaxone (N=39)
Pain/Burning at Injection Site (General disorders) | 1 (1) | 2 (2) — Complained of pain and/or burning at site of injection.
Headache/Dizziness (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 3 (4) — Back pain, pain in upper arm/shoulder above IN, neck/shoulder pain, shoulder pain, and pain in left arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No